CLINICAL TRIAL: NCT05583201
Title: A Single-center, Open-label, Single-arm Clinical Study of the Safety and Efficacy of KD-496 CAR-T Therapy in Advanced NKG2DL+/CLDN18.2+ Solid Tumors
Brief Title: NKG2D/CLDN18.2 CAR-T(KD-496) in the Treatment of Advanced NKG2DL+/CLDN18.2+ Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: jianming xu (Other)
Collaborators: KAEDI (Other)
Responsible Party: Sponsor-Investigator, jianming xu, Leading Site Principal Investigator, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Organization: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD-496-XJM
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer; Pancreatic Cancer; Solid Tumor
Keywords: NKG2D; CLDN18.2
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KD-496 cell infusion (Experimental): Each subject will receive KD-496 cell infusion
  Interventions: Biological: KD-496

INTERVENTIONS:
Biological: KD-496 — Autologous genetically modified anti-NKG2DL/CLDN18.2 CAR transduced T cells

SUMMARY:
This is a Phase 1, single-arm, single-center, open-label study to evaluate the safety and effectiveness of NKG2D/CLDN18.2-based CAR-T cells infusion in the treatment of advanced NKG2DL+/CLDN18.2+ solid tumors.

DETAILED DESCRIPTION:
This is an open-label, dose escalation/expansion study to assess the safety,tolerability, and efficacy of KD-496 cell infusion in patients with advanced NKG2DL+/CLDN18.2+ solid tumors. In this study, the enrollment of the patients must meet the inclusion and exclusion criteria. All subjects will be undergo screening, pre-treatment (cell product preparation, lymphodepleting chemotherapy), treatment and follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as advanced solid tumors histopathologically or cytologically, such as gastric cancer and pancreatic cancer. 2. Patients fail standard treatment , or cannot tolerate standard treatment, or there is no standard treatment, the standard treatment recommendations refer to the latest version of the guidelines of the national comprehensive cancer network (NCCN) or the guidelines of the Chinese society of Clinical Oncology (CSCO); 3. Age 18-75 years; 4. ECOG score 0-1; 5. Expected survival ≥ 3 months; 6. Patients must meet coagulation parameters and have adequate peripheral venous access for apheresis, and must also have enough PBMC to manufacture CAR T cells; 7. NKG2DL/CLDN18.2 (according to the positive comprehensive score of 0-12 points, positive SCORE of NKG2DL and CLDN18.2 ≥5) positive confirmed by Immunohistochemistry. Biopsy tissue must be no more than 2 year, if not, must obtain new tissue material from a recent surgical or diagnostic biopsy; 8. Eligible organ and bone marrow functions defined as follows:

1. Absolute neutrophil count ≥1.5×10^9/L, lymphocyte count ≥0.5×10^9/ L, platelet count ≥90×10^9/L, hemoglobin ≥90g/L (no blood transfusion or Erythropoietin within 7 days);
2. Total bilirubin ≤1.5ULN; (Patients with Gilbert syndrome were diagnosed with total bilirubin ≤3mg/dL) Serum alanineamino transferase (ALT) or aspartate aminotransferase(AST)≤3ULN(ALT and AST in patients with liver metastases ≤5ULN);
3. Creatinine ≤1.5ULN or eGFR≥60mL /min（Cockcroft and Gault）
4. International normalized ratio (INR) ≤1.2;
5. Lung function: ≤ grade 1 dyspnea(according to NCI-CTCAE V5.0), SaO2≥91%;
6. Cardiac function:

Cardiac ejection fraction (LVEF) detected by echocardiography or MUGA ≥50% 1 month before enrollment. 9. Patients must have measurable lesions as defined by RECIST 1.1; 10. If the patient is HBsAg positive or HBcAb positive, HBV-DNA should be < 2000IU/ml. HBsAg positive patients.Antiviral therapy must be received according to the Chronic Hepatitis B Prevention and Treatment Guidelines 2019.

11.Patients fully understand the test and voluntarily sign the informed consent; 12. Patient agree to use approved contraceptive methods (e.g., birth control pills, barrier devices, iuds, contraindicated drugs) during the study and for at least 13 months after last cell infusion, until no CAR-T cells were detected by two consecutive PCR tests.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV), Active hepatitis B (HBV DNA≥500IU/ml) or hepatitis c (anti-HCV positive and HCV RNA higher than the detection limit of analysis method)；
2. Patients had received any gene therapy (including CAR-T cell therapy) or any T cell therapy；
3. Patients had participated in other drug trials within 4 weeks prior to the study；
4. Patients with history or CT examination revealed active tuberculosis infection within 1 year before enrollment or patients diagnosed with active pulmonary tuberculosis 1 year ago without regular treatment；
5. Patients with sudden pulmonary disease, interstitial lung disease, pulmonary fibrosis, acute pulmonary disease, etc;
6. Subjects with pre-existing or active autoimmune diseases, or those with potential for recurrence (e.g., Wolf erythematosus systemic) Sores, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, kidneyGlomerulonephritis, etc.), or patients at high risk (such as those who have received organ transplants and require immunosuppressive therapy). But allowSubjects with the following diseases were enrolled:

1)Type 1 diabetic patients with stable disease after a fixed dose of insulin; 2)Only autoimmune hypothyroidism on hormone replacement therapy 3)Skin conditions that do not require systemic treatment (e.g., eczema, a rash of up to 10% of the body surface, silver flakes without ophthalmic symptoms Disease,etc.); 4)The use of immunosuppressants, such as steroids, should be phased out before the study begins if the patient has adrenal glands.If they are not functional, corticosteroids can be continued to replace the physiological dose (dose equivalent to ≤10 mg prednisone/day) 7.A history of severe heart disease, including medically poorly controlled hypertension (systolic blood pressure >160mmHg and/or diastolic blood pressure) Pressure >90mmHg), and any of the following conditions occurring within the past 6 months: patients with QT prolongation syndrome, screening,Phase 12 lead ECG results QTc interval >470mSEC, congestive heart failure (New York Heart Association grade ≥Class Ⅲ), cardiac angioplasty and stenting, myocardial infarction, unstable angina pectoris, severe arrhythmia or the researcher assessed heart disease that was not eligible for enrollment.

8. Clinically symptomatic brain metastases with the exception of patients with stable, asymptomatic brain metastases treated with radiotherapy or surgery for 14 days.

9. Other central nervous system disorders judged by the investigators to be likely to affect the trial: such as epilepsy/seizures, cerebral ischemia/hemorrhage, Dementia, cerebellar disease or autoimmune disease affecting the central nervous system.

10.Complicating hematologic malignancy or other primary malignant solid tumors, except in the following cases: 1) Patients with cervical or breast cancer accepted radical therapy without evidence of disease for more than 3 years; 2) The orthotopic tumor was successfully removed without definite resection patients with ≥5 years of evidence of disease.

11.Prior to apheresis, he received the following antitumor treatments:

1. Cytotoxic treatment within 14 days;
2. have received small molecule targeted therapy within 14 days or at least 5 half-lives, whichever is shorter,Therapy or investigational drug therapy, or treatment with invasive investigational medical devices;
3. Treatment with monoclonal antibodies within 21 days;
4. Immunomodulator therapy within 7 days;
5. Radiotherapy within 14 days. 12. Female subjects who are pregnant or breastfeeding during the screening period; 13. With a history of severe hypersensitivity to the primary therapeutic agents used in this study included fludarabine, cyclophosphamide, and PROPHYlaxis during pretreatment Tocilizumab and anti-infective drugs for CRS) 14.Untreated brain metastases or symptoms of brain metastases. 15.Patients with heart disease or poorly controlled high blood pressure who need treatment.

16.Patients with unstable or active peptic ulcers or gastrointestinal bleeding. 17.Patients who have a history of organ transplantation or are preparing for organ transplantation.

18.Patients requiring anticoagulant therapy (e.g., warfarin or heparin). 19.Patients requiring long-term antiplatelet therapy (aspirin,dose>300mg/d;clopidogrel,dose>75mg/d) 20.Patients had undergone major surgery or serious injury 4 weeks before the start of the study, or would undergo major surgery during the study.

21.Toxicity > grade 1 from previous antineoplastic therapy before screening (except alopecia).

22.Conditions that other researchers deemed inappropriate for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
treatment-emergent adverse events(TEAEs) | 3 months after single infusion
  An adverse event is any undesirable experience associated with the use of a medical product in a patient
Dose-limiting toxicity (DLT) rate | 3 months after single infusion
  A drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose.
CAR positive T cells in patients | 6 months after single infusion
  The time of CAR-T cell reach the peak and turn back to baseline

SECONDARY OUTCOMES:
Objective response rate(ORR) | 1 month, 2 month, 3 month, 6 month, 1 year after cell infusion
  objective tumor response rate will be calculated for patients with measurable disease per RECIST 1.1
Progression free survival(PFS) | 1 month, 2 month, 3 month, 6 month, 1 year after cell infusion
  the time from the date of first infusion of the KD-496 to the first documented disease progression (according to RECIST 1.1) or death (due to any cause), whichever occurs first
Complete remission (CR) | 1 month, 2 month, 3 month, 6 month, 1 year after cell infusion
  the time from the date of first infusion of KD-496 to death of the subject

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No